CLINICAL TRIAL: NCT00445302
Title: A Phase I Study Of The Safety, Pharmacokinetics, And Hematological Activity Of AMD3100 (240 µg/kg) In Subjects With Renal Impairment
Brief Title: Safety, Pharmacokinetics (PK), And Hematological Activity Of AMD3100 (Plerixafor) In Subjects With Renal Impairment
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Genzyme, a Sanofi Company (Industry)
Responsible Party: Medical Monitor, Genzyme
Organization: Sanofi (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AMD31001101
Record Dates: First submitted 2007-03-07; First posted 2007-03-08 (Estimated); Results first posted 2011-01-12 (Estimated); Last update posted 2014-03-13 (Estimated); Status verified 2014-02

CONDITIONS: Renal Impairment
Keywords: AMD3100
MeSH Terms: conditions — Renal Insufficiency | interventions — plerixafor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Normal renal function (Active Comparator): Participants with normal renal function (creatinine clearance (CLcr) > 90 ml/min) who serve as the study control. Participants treated with one dose of plerixafor (240 µg/kg) administered by subcutaneous (SC) injection.
  Interventions: Drug: plerixafor
- Mild renal impairment (Experimental): Participants have mild renal impairment (creatinine clearance (CLcr) = 51 to 80 mL/min). Participants treated with one dose of plerixafor (240 µg/kg) administered by subcutaneous (SC) injection.
  Interventions: Drug: plerixafor
- Moderate renal impairment (Experimental): Participants have moderate renal impairment (creatinine clearance (CLcr) = 31 to 50 mL/min). Participants treated with one dose of plerixafor (240 µg/kg) administered by subcutaneous (SC) injection.
  Interventions: Drug: plerixafor
- Severe renal impairment (Experimental): Participants have severe renal impairment (creatinine clearance (CLcr) < 31 mL/min, not requiring dialysis). Participants treated with one dose of plerixafor (240 µg/kg) administered by subcutaneous (SC) injection.
  Interventions: Drug: plerixafor

INTERVENTIONS:
Drug: plerixafor — Single dose of plerixafor (240 µg/kg) administered by subcutaneous (SC) injection
  Other Names: Mozobil; AMD3100

SUMMARY:
Eligible male and female subjects with renal impairment (aged 18-78 years) and healthy control subjects (aged 35 to 78 years) will be enrolled in the study. Subjects with renal impairment will be enrolled and entered into three groups based on their renal function: Mild Impairment, Moderate Impairment, and Severe Impairment(not requiring dialysis). Control subjects will have normal renal function.

The screening visits will occur within 14 days prior to plerixafor administration on study day one. Subjects will be monitored for 10 hours following administration of the study drug. In addition, subjects will return to the clinic at 24 and 48 hours after plerixafor administration for blood samples and safety assessments.

DETAILED DESCRIPTION:
This is a phase I, open label, multi-center study in which up to eighteen subjects with renal impairment and six healthy control subjects with normal renal function will receive a single dose of plerixafor (240 µg/kg) administered by subcutaneous (SC) injection.

Eligible male and female subjects with renal impairment (aged 18-78 years) and healthy control subjects (aged in the upper age range of the renal impairment subjects) will be enrolled in the study. Subjects with renal impairment will be enrolled and stratified into three cohorts using their Screening 24 hour urine collection to measured creatinine clearance (CLcr) values (an estimate of Glomerular Filtration Rate): Mild Impairment (CLcr = 51-80 ml/min), Moderate Impairment (CLcr = 31-50 ml/min), and Severe Impairment (CLcr <31 ml/min, not requiring dialysis). Control subjects will have normal renal function (CLcr >90 ml/min), as determined by a Screening 24 hour urine collection.

The screening visits will occur within 14 days prior to plerixafor administration on study day one. Subjects will be monitored for 10 hours following administration of the study drug. In addition, subjects will return to the clinic at 24 and 48 hours after plerixafor administration for blood samples and safety assessments.

This study was previously posted by AnorMED, Inc. In November 2006, AnorMED, Inc. was acquired by Genzyme Corporation. Genzyme Corporation is the sponsor of the trial.

ELIGIBILITY:
Inclusion Criteria:

* Signed patient informed consent form prior to any study procedures at Screening.
* Subject has not consumed alcohol in the 48 hours prior to the administration of study drug.
* Subject agrees to refrain from consumption of alcohol for the duration of the trial.
* Subject agrees to practice an approved method of contraception for the duration of the study.
* White blood cell count ≧3.5*10^9/L.
* Absolute polymorphonuclear leukocyte count >2.5*10^9/L.
* Platelet count >125*10^9/L.
* Serum glutamic oxaloacetic transaminase (SGOT), serum glutamic pyruvic transaminase (SGPT) and total bilirubin <2 times upper limit of normal (ULN).
* Negative for Human Immunodeficiency Virus (HIV).
* Age: Renal impairment subjects, 18-78 years. Control subjects, 35-78 years.
* Creatinine clearance measured from 24-hour urine collection (CLcr u): Renal impairment cohorts, Mild Impairment (CLcr u = 51-80 ml/min), Moderate Impairment (CLcr u = 31-50 ml/min), and Severe Impairment (CLcr u <31 ml/min, not requiring dialysis). Control subjects, CLcr u >90 ml/min.

Exclusion Criteria:

* Known sensitivity to plerixafor or any of its components.
* Pregnant or breast-feeding.
* Actual body weight exceeds 175% of ideal body mass index.
* Subjects judged by the investigator to be at significant risk of failing to comply with the requirements of the protocol.
* Any subject who has started new medication within 14 days prior to study drug administration.
* Treatment with an investigational product within 30 days prior to trial entry.
* Any significant untreated or newly diagnosed medical condition other than renal impairment that in the opinion of the investigator may interfere with the conduct of the study.
* Abnormal electrocardiogram with clinically significant rhythm disturbance,(ventricular arrhythmias), or other conduction abnormality that in the opinion of the investigator warrants exclusion of the subject from the trial.
* History of clinically significant thrombocytopenia.
* Received blood transfusions within 30 days prior to trial entry.
* Any subject who requires therapeutic intervention within the 30 days prior to administration of study medication in order to meet the inclusion/exclusion criteria.
* Active malignant/neoplastic disease requiring treatment of any kind.
* Active infection requiring antibiotics
* Renal impairment requiring any method of dialysis
* History of kidney transplant
* Subjects having clinical status or laboratory parameter deterioration between the time of enrollment and dosing with plerixafor (such that they no longer meet entry criteria) may be removed from the study at the discretion of the treating physician, principal investigator, or sponsor.

Ages: 18 Years to 78 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2006-01; Primary Completion 2007-08 (Actual); Study Completion 2007-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Genzyme, a Sanofi Company
Locations (3):
- United States (3):
  - Apex Research of Riverside, Santa Ana, California
  - Prism Research, 1000 Westgate Dr. suite 149, Saint Paul, Minnesota
  - Creighton University Medical Center, Omaha, Nebraska

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Cohort enrollment into the study was staged based on baseline creatinine clearance levels, with moderate renal impairment and control participants enrolled first. Severe renal impairment were enrolled following completion of the moderate renal impairment. Participants with mild renal impairment were enrolled last.
Groups:
- Normal Renal Function: Participants with normal renal function (creatinine clearance (CLcr) > 90 ml/min) used as a control. Participants treated with one dose of plerixafor (240 µg/kg) administered by subcutaneous (SC) injection.
- Mild Renal Impairment: Participants with mild renal impairment (CLcr = 51 to 80 mL/min). Participants treated with one dose of plerixafor (240 µg/kg) administered by subcutaneous (SC) injection.
- Moderate Renal Impairment: Participants with moderate renal impairment (CLcr = 31 to 50 mL/min). Participants treated with one dose of plerixafor (240 µg/kg) administered by subcutaneous (SC) injection.
- Severe Renal Impairment: Participants with severe renal impairment (CLcr < 31 mL/min, not requiring dialysis). Participants treated with one dose of plerixafor (240 µg/kg) administered by subcutaneous (SC) injection.
Period: Overall Study
Arm/Group | Normal Renal Function | Mild Renal Impairment | Moderate Renal Impairment | Severe Renal Impairment
Started | 6 | 5 | 6 | 6
Completed | 6 | 5 | 6 | 6
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Normal Renal Function | Mild Renal Impairment | Moderate Renal Impairment | Severe Renal Impairment | Total
Number analyzed (Participants) | 6 | 5 | 6 | 6 | 23
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.3 (5.50) | 56.2 (14.45) | 65.0 (5.83) | 55.7 (11.98) | 54.7 (12.51)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 2 | 4 | 11
  Male | 4 | 2 | 4 | 2 | 12
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 1 | 3 | 3 | 5 | 12
  African-American | 4 | 1 | 2 | 1 | 8
  Hispanic/Latino | 1 | 1 | 1 | 0 | 3

OUTCOME MEASURES:

1. Primary Outcome: Dose-Normalized Maximum Concentration of Plerixafor (Cmax)
Description: Evaluation of Cmax following a single dose of 240 µg/kg plerixafor administered on Day 1. Cmax was normalized by dose.
Time Frame: Pre-dose of plerixafor to 24 hours post-plerixafor
Population: Intent-to-treat population
Measure: Mean (Standard Deviation); unit: ng/mL/ug
Arm/Group | Normal Renal Function | Mild Renal Impairment | Moderate Renal Impairment | Severe Renal Impairment
Number analyzed (Participants) | 6 | 5 | 6 | 6
ng/mL/ug | 0.0452 (0.0145) [60.03 to 96.90] | 0.0388 (0.0095) [74.13 to 117.02] | 0.0490 (0.0150) [69.56 to 109.81] | 0.0475 (0.0110)
Statistical Analysis 1: Comparison: Normal Renal Function vs Mild Renal Impairment; Test type: Superiority or Other; Ratio of least squares means (%) = 87.09, 90% CI 2-sided [63.59 to 119.26]
Statistical Analysis 2: Comparison: Normal Renal Function vs Moderate Renal Impairment; Test type: Superiority or Other; Ratio of least squares means(%) = 106.60, 90% CI [78.99 to 143.87]
Statistical Analysis 3: Comparison: Normal Renal Function vs Severe Renal Impairment; Test type: Superiority or Other; Ratio of least squares means (%) = 106.76, 90% CI [79.11 to 144.08]

2. Secondary Outcome: Change From Baseline in Absolute CD34+ Cell Counts at Day 2
Description: Change in circulating CD34+ cells from baseline to Day 2 (24 hours post-plerixafor) following a single dose of plerixafor. Change from baseline = CD34+ cell count at 24 hours post dose - CD34+ cell count at Baseline.
Time Frame: Baseline, Day 2
Population: An intent-to-treat approach was used to calculate the outcome measure in each arm/group.
Measure: Mean (Standard Deviation); unit: cells/mm^3
Arm/Group | Normal Renal Function | Mild Renal Impairment | Moderate Renal Impairment | Severe Renal Impairment
Number analyzed (Participants) | 6 | 5 | 6 | 6
cells/mm^3 | 10.5 (6.19) | 11.8 (2.49) | 14.3 (14.24) | 23.0 (18.20)

3. Secondary Outcome: Change From Baseline in Absolute White Blood Cell (WBC) Counts at Day 2
Description: Change in absolute white blood cells from baseline to Day 2 (24 hours post-plerixafor) following a single dose of plerixafor. Change from baseline = absolute white blood cells at 24 hours post dose - absolute white blood cells at Baseline.
Time Frame: Baseline and Day 2
Population: An intent-to-treat approach was used to calculate the outcome measure in each arm/group.
Measure: Mean (Standard Deviation); unit: cells/mm^3
Arm/Group | Normal Renal Function | Mild Renal Impairment | Moderate Renal Impairment | Severe Renal Impairment
Number analyzed (Participants) | 6 | 5 | 6 | 6
cells/mm^3 | 7416.7 (1986.37) | 10540.0 (2785.32) | 12133.3 (4501.41) | 14975.0 (5030.82)

4. Primary Outcome: Dose-Normalized Area Under the Plerixafor Concentration Time Curve From Time 0 to 24 Hours Post-dose (AUC0-24h)
Description: Evaluation of AUC0-24 hour following a single dose of 240 µg/kg plerixafor administered on Day 1. AUC0-24 was normalized by dose.
Time Frame: Pre-dose of plerixafor to 24 hours post-plerixafor
Population: Intent-to-treat population
Measure: Mean (Standard Deviation); unit: hr*ng/mL/ug
Arm/Group | Normal Renal Function | Mild Renal Impairment | Moderate Renal Impairment | Severe Renal Impairment
Number analyzed (Participants) | 6 | 5 | 6 | 6
hr*ng/mL/ug | 0.2277 (0.0360) | 0.2866 (0.0854) | 0.3550 (0.0965) | 0.3872 (0.0688)
Statistical Analysis 1: Comparison: Normal Renal Function vs Mild Renal Impairment; Test type: Superiority or Other; Ratio of least squares means (%) = 121.74, 90% CI [91.86 to 161.43]
Statistical Analysis 2: Comparison: Normal Renal Function vs Moderate Renal Impairment; Test type: Superiority or Other; Ratio of least squares means (%) = 151.44, 90% CI [115.78 to 198.09]
Statistical Analysis 3: Comparison: Normal Renal Function vs Severe Renal Impairment; Test type: Superiority or Other; Ratio of least squares means (%) = 169.51, 90% CI [129.59 to 221.72]

5. Secondary Outcome: Number of Participants in Overall Safety Summary of Adverse Events (TEAE)
Description: Number of participants with adverse events (AEs) collected from Day 1 (post plerixafor administration) to Day 3. AEs were graded by the investigator using the World Health Organization (WHO) Adverse Event Grading Scale and were assessed for severity (mild, moderate, severe, life-threatening) and relatedness to study treatment (5 point scale from 'not related' to 'definitely related').
Time Frame: up to Day 3
Population: The safety analyses were performed on the Safety Population which consisted of all subjects who received plerixafor.
Measure: Number; unit: participants
Arm/Group | Normal Renal Function | Mild Renal Impairment | Moderate Renal Impairment | Severe Renal Impairment
Number analyzed (Participants) | 6 | 5 | 6 | 6
participants
  AE Severity (Mild) | 3 | 1 | 3 | 2
  AE Severity (Moderate) | 2 | 1 | 1 | 2
  AE Severity (Severe) | 0 | 0 | 0 | 0
  AE Severity (Life Threatening) | 0 | 0 | 0 | 0
  AE Relationship to Drug (Definitely related) | 4 | 2 | 2 | 2
  AE Relationship to Drug (Probably related) | 1 | 0 | 2 | 0
  AE Relationship to Drug (Possibly related) | 0 | 0 | 0 | 2
  AE Relationship to Drug (Probably not related) | 0 | 0 | 0 | 0
  AE Relationship to Drug (Definitely not related) | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: From the time of the first dose of plerixafor to study Day 3 (study completion).
Description: In the event a single participant has experienced both a serious and a non-serious form of the same adverse event term, the individual has been included in the numerator ("number of affected participants") of both adverse event tables.
  Each AE table includes events, regardless of reported relationship to study treatment or grade.
Arm/Group | Normal Renal Function | Mild Renal Impairment | Moderate Renal Impairment | Severe Renal Impairment
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/5 | 0/6
Other Adverse Events (participants affected / at risk) | 4/6 | 4/6 | 2/5 | 5/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Normal Renal Function (N=6) | Mild Renal Impairment (N=6) | Moderate Renal Impairment (N=5) | Severe Renal Impairment (N=6)
Leukocytosis (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 — This event of leukocytosis reflects a white blood cell (WBC) count of 26.44*10^9/L.
Abdominal distension (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 0 | 2 | 2
Hypoaesthesia oral (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 1 | 0 | 2
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Feeling hot (General disorders) | 0 | 0 | 1 | 0
Injection site bruising (General disorders) | 0 | 1 | 0 | 0
Injection site erythema (General disorders) | 1 | 1 | 1 | 2
Injection site rash (General disorders) | 0 | 0 | 1 | 0
Injection site reaction (General disorders) | 1 | 0 | 1 | 1
Red blood cells urine positive (Investigations) | 1 | 0 | 0 | 0
Urinary sediment present (Investigations) | 1 | 0 | 0 | 0
Urine analysis abnormal (Investigations) | 1 | 0 | 0 | 0
White blood cell count increased (Investigations) | 0 | 1 | 0 | 0
White blood cells urine positive (Investigations) | 1 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 2
Dizziness (Nervous system disorders) | 0 | 0 | 1 | 1
Dysgeusia (Nervous system disorders) | 0 | 1 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 0 | 1
Paraesthesia (Nervous system disorders) | 2 | 0 | 1 | 1
Sinus headache (Nervous system disorders) | 0 | 0 | 1 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 1 | 0
Hyperventilation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Flushing (Vascular disorders) | 1 | 0 | 0 | 2
Phlebitis (Vascular disorders) | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
In multi-site studies, PI can publish after Genzyme publishes or 12 months after study completion. PI gives Genzyme a draft 30 days before publication. Genzyme can ask that confidential information be removed, and can defer publication another 90 days upon notifying PI that it will file a patent application on inventions contained in the draft.